CLINICAL TRIAL: NCT05212246
Title: CSP #2019 - Basal Cell Carcinoma Chemoprevention Trial (B3C)
Brief Title: Basal Cell Carcinoma Chemoprevention Trial
Acronym: B3C
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2019
Record Dates: First submitted 2022-01-14; First posted 2022-01-28 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Basal Cell Carcinoma
Keywords: Basal Cell Carcinoma; chemoprevention; imiquimod; facial skin cancer; skin cancer prevention; squamous cell carcinoma; keratinocyte carcinoma; actinic keratosis; quality of life; side effects; treatment compliance; automated text messaging; cost comparison and cost effectiveness; implementation science
MeSH Terms: conditions — Carcinoma, Basal Cell; Carcinoma, Squamous Cell; Keratosis, Actinic; Patient Compliance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 5% Imiquimod Cream (Experimental): Topical 5% Imiquimod cream will be applied once daily to the face in a thin layer for 12 weeks. Three packets of cream will be defined as one dose or application. The cream should be applied to the face prior to normal sleeping hours (it is readily absorbed) and left on the skin for 6-10 hours (i.e. overnight). Rest periods will be allowed if bothersome side effects occur.
  Interventions: Drug: 5% Imiquimod cream
- Placebo Vehicle Control Cream (Placebo Comparator): The placebo vehicle control cream will be a virtually identical cream (to the Imiquimod cream) that contains no Imiquimod. This cream will be applied once daily to the face in a thin layer for 12 weeks. Three packets of cream will be defined as one dose or application. The cream should be applied to the face prior to normal sleeping hours (it is readily absorbed) and left on the skin for 6-10 hours (i.e. overnight). Rest periods will be allowed if bothersome side effects occur.
  Interventions: Drug: Placebo Vehicle Control Cream

INTERVENTIONS:
Drug: 5% Imiquimod cream — Topical 5% Imiquimod cream will be applied once daily to the face in a thin layer for 12 weeks. Three packets of cream will be defined as one dose or application. The cream should be applied to the face prior to normal sleeping hours (it is readily absorbed) and left on the skin for 6-10 hours (i.e. overnight). Rest periods will be allowed if bothersome side effects occur.
  Other Names: IMQ
  Arms: 5% Imiquimod Cream
Drug: Placebo Vehicle Control Cream — The placebo vehicle control cream will be a virtually identical cream (to the Imiquimod cream) that contains no Imiquimod. This cream will be applied once daily to the face in a thin layer for 12 weeks. Three packets of cream will be defined as one dose or application. The cream should be applied to the face prior to normal sleeping hours (it is readily absorbed) and left on the skin for 6-10 hours (i.e. overnight). Rest periods will be allowed if bothersome side effects occur.
  Other Names: Placebo
  Arms: Placebo Vehicle Control Cream

SUMMARY:
This is an intent-to-treat, parallel design, multicenter randomized trial and the primary intervention is a double-blind comparison of Imiquimod (IMQ) vs. placebo cream for preventing basal cell carcinoma (BCC) of the skin on the face at one year and over 3 years after therapy. Participants will apply the IMQ or placebo cream to the face daily at bedtime for 12 weeks. This study will recruit 1630 Veterans at high risk of BCC from 17 VA medical centers.

DETAILED DESCRIPTION:
Basal Cell Carcinoma (BCC) is the most common cancer in the United States. It afflicts 2 to 3 million Americans each year, more than all non-skin cancers combined. Notably, US active duty military and Veterans are at higher risk for developing BCC, with at least 49,000 Veterans treated for the disease in 2010. BCC usually occurs on the face and hence can result in high morbidity and disfigurement with substantial associated expense both in the overall population (estimated at $3 billion in 2013), and among Veterans (estimated at $86 million in 2012) served by Veterans Health Administration (VHA). Morbidity and disfigurement are particularly important due to their impact on key facial structures (e.g. eyelids, nose, etc). After BCC diagnosis, subsequent monitoring for BCC (ex. return specialist visits for dermatologic examinations) and treatments following diagnosis (surgeries most commonly, but also radiation therapy or chemotherapy) significantly contribute to healthcare costs. This large incidence, morbidity, and cost could potentially be minimized through preventative measures, but currently there are no treatment options for preventing BCC.

The primary goal of this study is to investigate the efficacy of topical Imiquimod (IMQ) for the prevention of BCC. IMQ, a topical immunostimulatory medication with a very low rate of side effects, is potentially capable of meeting this need. IMQ is already FDA approved as a safe and effective treatment for superficial BCC, as well as for actinic keratosis and nodular BCC. The investigators have reason to suspect that IMQ may also be able to prevent the occurrence of BCC or to destroy clinically-unrecognized precursors of BCC, thereby reducing the risk of BCC development.

CSP #2019 is an intent-to-treat, double-blind, parallel design, multicenter randomized trial of IMQ vs. placebo cream for preventing BCC on the face at one year and over 3 years after therapy. Nine out of 17 participating centers will start recruitment in the first year of the study (Phase 1 centers), with 5 centers randomly assigned to offer daily study treatment reminders via the Annie app and the other 4 centers not offering it. The remaining 8 centers (Phase 2 centers) will start in the second year of the study, with half of the centers randomized to offer daily study treatment reminders via the Annie app and the other half not offering it. Participants in each center will be randomly allocated (1:1) to either topical IMQ or placebo (vehicle control cream). Study participants, staff and study dermatologists will not know which treatment the participant receives. Participants will apply IMQ or placebo cream to the face daily at bedtime for a total of 12 weeks. In-person visits will occur at weeks 6 and 12 during treatment, and at months 6, 12, 18, 24, 30, and 36 during active follow-up to assess study outcomes. Full skin exams will be performed and other outcome data collected at every scheduled in-person visit with the exception that only facial skin exams are performed at weeks 6 and 12 visits. Telephone interviews will occur every week through week 13 (other than weeks 6 and 12, due to an in-person visit), as well as at months 9, 15, 21, 27, and 33. Follow-up will include 3 years of active follow-up with participants, followed by 1 year of passive follow-up during which study outcome information will only be captured from medical records.

ELIGIBILITY:
Inclusion Criteria:

* Veteran age 18 years or older
* 2 (or more) qualifying BCC lesions in the prior 5 years, with at least one located on the face, neck, ears, or scalp. "Qualifying lesions are those that meet the two inclusion criterion bullet points below, and none of the exclusion criteria listed in "B".
* Qualifying lesions not in a field of prior radiation therapy.
* Qualifying lesions not a recurrence after treatment, but the original lesion can qualify whether it recurred or not.

Exclusion Criteria:

* AK or KC field therapy on the face (5-FU cream, IMQ, diclofenac gel, chemical peel, or photodynamic therapy) for BCC treatment on the face in the last 2 months because it can cause inflammation that may interfere with the IMQ treatment. After 2 months, these patients can be included.
* IMQ therapy on the face in the past year, although such therapy in the more distant past is not an exclusion.
* Suspicious skin lesions suggestive of any type of skin cancer present on the face at the initial exam conducted for the study must be removed and have another skin exam to confirm the facial skin cancer is cleared for 1 month prior to randomization so that the investigators can be confident that skin cancer lesions that arise during the trial are new.
* Currently receiving or received in the past two months: immune checkpoint inhibitor, hedgehog pathway inhibitor, or oral capecitabine.
* History of cutaneous T-cell lymphoma within the past year, but low-grade prostate cancer, patch stage CTCL, breast cancer, and history of solid hematologic cancer deemed to be in remission will be included.
* Genetic disorder associated with very high basal cell skin cancer risk (i.e., basal cell nevus syndrome, xeroderma pigmentosum) because prevention efforts with IMQ may have dramatically different efficacy in these patients compared to the general high-risk population.
* Solid organ or bone marrow transplant recipient such as renal, hepatic, or cardiac transplant because these patients are at increased risk of KC (much greater risk of SCC than BCC) and the associated immunodeficiency may affect the effectiveness of IMQ
* Radiation therapy to the face
* Known allergy to IMQ or cream vehicle
* Woman currently pregnant or breast feeding
* Woman of childbearing potential unwilling to use birth control
* Judged by investigator to have a very high mortality risk within a year due to co-morbid illness
* Judged by investigator to be unlikely to comply with protocol requirements
* Judged by investigator not to be competent to provide informed consent
* Unable to communicate in English
* Enrolled in another therapeutic interventional trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1630 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2032-05-03 (Estimated); Study Completion 2032-05-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with a new Basal Cell Carcinoma (BCC) on the face at 1 year | 1 year from the time of randomization
  Skin exams will occur at baseline and at 6-month intervals after study randomization. Diagnosis of a new BCC will be ascertained by a biopsy under local anesthesia in an outpatient setting, as is the standard of care. Every biopsy performed on the face of a participant during the trial will be processed per standard clinical operating procedures, as determined by their blinded clinician for the purposes of patient management. The biopsy will be sent for reading by a blinded central dermatopathologist with known high reliability (intra-rater and inter-rater with two other board-certified dermatopathologists) for diagnosing BCC. This central dermatopathologist diagnosis will be used for study purposes. Skin cancers diagnosed outside of the VA, and associated surgeries, will be systematically sought in all participants by participant interview and review of medical records to ensure that the outcome measure is complete.
Basal Cell Carcinoma (BCC) free time to a new BCC on the face over 3 years | 3 years from the time of randomization
  Basal Cell Carcinoma (BCC) free time to a new BCC on the face over 3 years is defined as the time in years from treatment randomization to the first occurrence of a new BCC on the face. Participants who do not develop a new BCC on the face by 3 years will be considered censored observations. Skin exams will occur at baseline and at 6-month intervals after study randomization.

SECONDARY OUTCOMES:
Proportion of participants with a new Squamous Cell Carcinoma (SCC) on the face at 1 year | 1 year from the time of randomization
  Diagnosis of a new SCC will be ascertained by a biopsy under local anesthesia in an outpatient setting, as is the standard of care. Every biopsy performed on the face of a participant during the trial will be processed per standard clinical operating procedures, as determined by their blinded clinician for the purposes of patient management, and the biopsy will also be sent for reading by a blinded central dermatopathologist with known high reliability (intra-rater and inter-rater with two other board-certified dermatopathologists) for diagnosing SCC. This central dermatopathologist diagnosis will be used for study purposes. Skin cancers diagnosed outside of the VA, and associated surgeries, will be systematically sought in all participants by participant interview and review of medical records to ensure that the outcome measure is complete.
Squamous Cell Carcinoma (SCC) free time to a new SCC on the face over 3 years | 3 years from the time of randomization
  Squamous Cell Carcinoma (SCC) free time to a new SCC on the face over 3 years is defined as the time in years from treatment randomization to the first occurrence of a new SCC on the face. Participants who do not develop a new SCC on the face by 3 years will be considered censored observations.
Total Actinic Keratosis (AK) reduction on the face over time during treatment and active follow-up | 3 years from the time of randomization
  AK reduction persistence over time will be assessed using total AK counts (on the face only) evaluated at in-person visits at weeks 6 and 12 and months 6, 12, 18, 24, 30, and 36, and will be analyzed as a repeated measures outcome.
AK reduction in each Olsen grade on the face over time during treatment and active follow-up | 3 year from the time of randomization
  AK reduction in each Olsen grade on the face over time will be assessed using AK counts (on the face only) in each Olsen grade evaluated at in-person visits at weeks 6 and 12 and months 6, 12, 18, 24, 30, and 36, and will be analyzed as a repeated measures outcome.
Proportion of participants with any facial Actinic Keratosis (AK) biopsies or surgical removal on the face at 1 year | 1 year from the time of randomization
  The proportion of participants with any facial Actinic Keratosis (AK) biopsies or surgical removal on the face from the start of study treatment up to 1 year. Data collection regarding AK biopsies on the face will be assessed at weeks 6 and 12 during treatment, and months 6, 9, and 12 during active follow-up.
Proportion of participants with a cheek or forehead primary Basal Cell Carcinoma (BCC) versus other areas of the face at 1 year | 1 year from the time of randomization
  Facial regions will be dichotomized to forehead and cheeks versus other areas include the ear, eye (including eyebrows), and nose areas. We will characterize subsites where BCC occurs and assess the effect of IMQ on preventing BCC on the forehead and cheek areas compared to elsewhere on the face.
Proportion of participants with a cheek or forehead primary Basal Cell Carcinoma (BCC) versus other areas of the face at 3 years | 3 years from the time of randomization
  Facial regions will be dichotomized to forehead and cheeks versus other areas include the ear, eye (including eyebrows), and nose areas. We will characterize subsites where BCC occurs and assess the effect of IMQ on preventing BCC on the forehead and cheek areas compared to elsewhere on the face.
Proportion of participants with a facial primary Basal Cell Carcinoma (BCC) of aggressive histologic subtypes at 1 year | 1 year from the time of randomization
  Higher risk histologic subtypes include infiltrative/morpheaform and nodular/infiltrative BCCs.
Proportion of participants with a facial primary Basal Cell Carcinoma (BCC) of aggressive histologic subtypes at 3 years | 3 years from the time of randomization
  Higher risk histologic subtypes include infiltrative/morpheaform and nodular/infiltrative BCCs.
Proportion of participants who have experienced a facial primary Basal Cell Carcinoma (BCC) of high severity at 1 year | 1 year from the time of randomization
  The proportion of participants who have experienced a facial primary Basal Cell Carcinoma (BCC) of high severity at 1 year will be determined. To be considered a high severity (i.e. high morbidity) BCC, the tumor must have at least moderate severity and of high severity one of the following features:
  i.AJCC stage 3 or 4 BCC ii.BCC requiring radiation iii.BCC requiring multidisciplinary surgery (i.e. oculoplastics, ENT, or neurosurgery, with or without concomitant Mohs micrographic surgery) iv.BCC requiring systemic treatment
Proportion of participants who have experienced a facial primary Basal Cell Carcinoma (BCC) of high severity at 3 years | 3 years from the time of randomization
  The proportion of participants who have experienced a high severity Basal Cell Carcinoma (BCC) at 3 years will be determined. To be considered a high severity (i.e. high morbidity) BCC, the tumor must have at least one of the following features:
  i.AJCC stage 3 or 4 BCC ii.BCC requiring radiation iii.BCC requiring multidisciplinary surgery (i.e. oculoplastics, ENT, or neurosurgery, with or without concomitant Mohs micrographic surgery) iv.BCC requiring systemic treatment
Proportion of participants who have experienced a high or moderate severity facial primary Basal Cell Carcinoma (BCC) at 1 year | 1 year from the time of randomization
  The proportion of participants who have experienced a high or moderate severity Basal Cell Carcinoma (BCC) at 1 year will be determined. To be considered a high severity (i.e. high morbidity) BCC, the tumor must have at least one of the following features:
  i.AJCC stage 3 or 4 BCC ii.BCC requiring radiation iii.BCC requiring multidisciplinary surgery (i.e. oculoplastics, ENT, or neurosurgery, with or without concomitant Mohs micrographic surgery) iv.BCC requiring systemic treatment
  To be considered a moderate severity (i.e. moderate morbidity) BCC, the tumor must require surgical removal, which may include removal with Mohs micrographic surgery, but not meet the criteria for high severity. To be included in mild severity/morbidity, the tumor must not require surgical intervention.
Proportion of participants who have experienced a high or moderate severity facial primary Basal Cell Carcinoma (BCC) at 3 years | 3 years from the time of randomization
  The proportion of participants who have experienced a high or moderate severity Basal Cell Carcinoma (BCC) at 3 years will be determined. To be considered a high severity (i.e. high morbidity) BCC, the tumor must have at least one of the following features:
  i.AJCC stage 3 or 4 BCC ii.BCC requiring radiation iii.BCC requiring multidisciplinary surgery (i.e. oculoplastics, ENT, or neurosurgery, with or without concomitant Mohs micrographic surgery) iv.BCC requiring systemic treatment
  To be considered a moderate severity (i.e. moderate morbidity) BCC, the tumor must require surgical removal, which may include removal with Mohs micrographic surgery, but not meet the criteria for high severity. To be included in mild severity/morbidity, the tumor must not require surgical intervention.
Proportion of participants with any side effect of treatment during the treatment phase (weeks 1-13) | Weeks 1-13 after randomization
  The proportion of participants with any side effect of treatment during the 12 weeks of the active treatment period or the week following the end of active treatment (week 13).
Proportion of participants not tolerating the side effects during the treatment phase | Weeks 12 after randomization
  Tolerability of treatment side effects will be assessed at the end of the treatment (week 12) and it will be a binary response (yes/no).
Facial photograph toxicity scores at week 6 and week 12 | Weeks 6 and 12 after randomization
  Photographs of the face will be taken at weeks 6 and 12 in-person visits and translated into a numerical score on the toxicity scale established and used in CSP #562 - the VA Keratinocyte Carcinoma Chemoprevention (VAKCC) Trial.
Skindex-16 quality of life scores at 12 weeks | Twelve weeks after randomization
  The Skindex-16 is a 16-item scale to measure the effects of skin disease on a patient's quality of life. All item responses are transformed to a linear scale of 100, varying from 0 (no effect) to 100 (effect experienced all the time). Skindex scores are reported as three scale scores corresponding to the following three domains or subscales: Symptom, Emotional, Functional. A scale score is the average of a patient's responses to items in a given domain. Higher domain scale scores represent worse quality of life.
Skindex-16 quality of life scores at 6 months | Six months after randomization
  The Skindex-16 is a 16-item scale to measure the effects of skin disease on a patient's quality of life. All item responses are transformed to a linear scale of 100, varying from 0 (no effect) to 100 (effect experienced all the time). Skindex scores are reported as three scale scores corresponding to the following three domains or subscales: Symptom, Emotional, Functional. A scale score is the average of a patient's responses to items in a given domain. Higher domain scale scores represent worse quality of life.
Functional Assessment of Cancer Therapy-General (FACT-G) Physical Well-being score at 12 weeks | Twelve weeks after randomization
  The Functional Assessment of Cancer Therapy - General (FACT-G) is a 27-item questionnaire designed to measure four domains of HRQOL in cancer patients: Physical, social, emotional, and functional well-being. Only the 7-item Physical Well-being subscale is being used in this study. The Physical Well-being score range is 0-28, and the higher score, the better the quality of life.
Functional Assessment of Cancer Therapy-General (FACT-G) Physical Well-being score at 6 months | Six months after randomization
  The Functional Assessment of Cancer Therapy - General (FACT-G) is a 27-item questionnaire designed to measure four domains of HRQOL in cancer patients: Physical, social, emotional, and functional well-being. Only the 7-item Physical Well-being subscale is being used in this study. The Physical Well-being score range is 0-28, and the higher score, the better the quality of life.
Proportion of participants indicating acceptability of the study treatment cream at 12 weeks | Twelve weeks after randomization
  The proportion of participants indicating acceptability of their assigned treatment cream at 12 weeks will be summarized by treatment group. Acceptability will be assessed by asking participants at 12 weeks whether they would be willing to use the cream they received again in the future if the cream is determined to be effective in reducing their risk of developing future skin cancer on the face.
Study treatment compliance status during the 12 weeks of active treatment by treatment group | Twelve weeks after randomization
  Medication compliance will be defined as a binary outcome (>=80% compliance vs <80% compliance). Individuals applying 67 or more of the expect 84 doses (67/84=80% with rounding) will be considered >=80% medication compliant, while those applying <67 doses will be considered <80% compliant.
Study treatment compliance status during the 12 weeks of active treatment by study site Annie application status | Twelve weeks after randomization
  Study treatment compliance status will be defined as a binary outcome (>=80% compliance vs <80% compliance). Individuals applying 67 or more of the expect 84 doses (67/84=80% with rounding) will be considered >=80% medication compliant, while those applying <67 doses will be considered <80% compliant.
  The US Department of Veterans Affairs has developed an automated text message service application called Annie that can send automated treatment reminders to Veterans if they register/enroll in Annie and consent to receive Annie text messages. Nine of the 17 study sites will be randomly selected to offer the Annie application to their study participants. The medication compliance status during the 12 weeks of active treatment (as defined above) will be presented for the 9 study sites offering the Annie app and the 8 sites not offering it (irrespective of study treatment group).
Study treatment compliance status during the 12 weeks of active treatment by Annie application status only at sites offering Annie | Twelve weeks after randomization
  Study treatment compliance status will be defined as a binary outcome (>=80% compliance vs <80% compliance). Individuals applying 67 or more of the expect 84 doses (67/84=80% with rounding) will be considered >=80% medication compliant, while those applying <67 doses will be considered <80% compliant.
  Veterans Affairs has developed an application called Annie that can send text treatment reminders to Veterans if they enroll in Annie. Nine of the 17 sites will be randomly selected to offer Annie to their participants. Annie use is voluntary and not required for participation. Among the sites offering Annie, we will ask participants whether they received any treatment reminders via Annie & a categorical Annie use variable will be created. Only for the 9 sites offering Annie, the medication compliance status (as defined above) will be presented for the participants that used Annie and those that didn't.
Proportion of participants with a new Basal Cell Carcinoma (BCC) on the face at 1 year by study treatment compliance status | One year after randomization
  Skin exams will occur at baseline & 6 months after randomization. Diagnosis of a new facial BCC will be via biopsy under local anesthesia in an outpatient setting (standard of care). Every facial biopsy will be processed per standard operating procedures, as determined by the blinded clinician for the purposes of patient management. Biopsies will be read by blinded central dermatopathologist with known high reliability (intra-rater & inter-rater with 2 board-certified dermatopathologists) for diagnosing BCC. Central dermatopathologist diagnosis will be used for study purposes. BCC diagnosed outside VA & surgeries will be collected by participant interview and review of medical records to ensure the outcome measure is complete. Medication compliance will be defined as a binary outcome (>=80% vs <80%). Individuals applying 67 or more of the expect 84 doses (67/84=80% with rounding) will be considered >=80% compliant, while those applying <67 doses will be considered <80% compliant.
Basal Cell Carcinoma (BCC) free time to a new BCC on the face over 3 years by study treatment compliance status | Three years from the time of randomization
  Basal Cell Carcinoma (BCC) free time to a new BCC on the face over 3 years is defined as the time in years from treatment randomization to the first occurrence of a new BCC on the face. Participants who do not develop a new BCC on the face by 3 years will be considered censored observations. Skin exams will occur at baseline and at 6-month intervals after study randomization.
  Medication compliance status will be defined as a binary outcome (>=80% compliance vs <80% compliance). Individuals applying 67 or more of the expect 84 doses (67/84=80% with rounding) will be considered >=80% medication compliant, while those applying <67 doses will be considered <80% compliant.

CONTACTS AND LOCATIONS:
Overall Officials: Martin A. Weinstock, MD, Study Chair — Providence VA Medical Center, Providence, RI
Locations (1):
- Providence VA Medical Center, Providence, RI, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
After the main results of this study have been published, de-identified data from the study may be shared with other VA investigators, other Federal health agencies, or academic institutions for additional analyses provided this use has been approved by CSP, the appropriate VA oversight committee(s), and there is an agreement in place that defines the limits of this use.
  With the participant's approval and as approved by local Institutional Review Boards (IRBs), deidentified study data will be moved into a data repository where other CSP studies are maintained after the study has ended. This data could be used for future research on the conditions, characteristics, complications, and treatments covered in the proposed work.
Supporting Information: Study Protocol, SAP
Time Frame: 10 years after primary publication